CLINICAL TRIAL: NCT04950582
Title: In Vitro Analysis of Human Urine With the CloudCath Device
Status: Suspended | Type: Observational
Why Stopped: temporary pause due to business priorities
Sponsor: CloudCath (Industry)
Responsible Party: Sponsor
Other Study IDs: CC-L-008
Record Dates: First submitted 2021-06-09; First posted 2021-07-06 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Urinary Tract Infections
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- UTI-high risk patients: patients who are at high risk for developing a urinary tract infection (UTI).
  Interventions: Diagnostic Test: Spectral characteristics assessment

INTERVENTIONS:
Diagnostic Test: Spectral characteristics assessment — Urine sample analysis for evidence of urinary tract infection

SUMMARY:
This is a multi-center feasibility study to assess the in vitro function of the CloudCath Device that is being developed to derive clinically-relevant information from the optical characteristics of urine.

DETAILED DESCRIPTION:
Specimens will be obtained from participants with indwelling catheters in hospital or home settings, who are suspected to be at high risk for urinary tract infection.

To evaluate the performance of the CloudCath Device in repeated measurements over time, multiple specimens may be obtained from the same patients over multiple days or months.

Each sample will be divided into multiple aliquots. One part will be analyzed using the CloudCath Device and reference devices. Another part may be submitted to an independent lab for standard analytical tests.

ELIGIBILITY:
Inclusion Criteria:

* provide a signed informed consent
* patient has an implanted urinary catheter (i.e., Foley, Texas, ureteral)

Exclusion Criteria:

* any condition that the investigator feels may confound the study results or place the participant at risk by participating in the study
* currently taking antibiotics for any reason other than for treatment of urinary tract infection (UTI)
* suprapubic bladder catheter implanted

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with indwelling urinary catheters
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-06-04 (Actual); Primary Completion 2024-06-15 (Estimated); Study Completion 2024-06-15 (Estimated)

PRIMARY OUTCOMES:
Spectral characteristics of urine specimens | During the period of time that the patient is catheterized (expected to be up to ~1 week)
  A quantitative analysis of the spectral properties of the urine specimen using a proprietary algorithm that results in a quantitative CloudCath Turbidity Score (0-100, with higher values indicating more turbidity).

CONTACTS AND LOCATIONS:
Overall Officials: Ben Briggs, MD, PhD, Study Director — University of California, San Francisco
Locations (1):
- CloudCath Investigational Site, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No